CLINICAL TRIAL: NCT02242383
Title: Morning Hypertension and Monitoring of Metabolism (AWB Morgenhochdruck & Stoffwechselmonitoring)
Brief Title: Evaluation of Efficacy and Tolerability of Micardis® / MicardisPlus® Under Usual Daily-practice Prescribing in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.485
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Essential hypertension
  Interventions: Drug: Telmisartan; Drug: Telmisartan in combination with hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan
Drug: Telmisartan in combination with hydrochlorothiazide

SUMMARY:
To evaluate efficacy and tolerability of Micardis® / MicardisPlus® under usual daily-practice prescribing conditions with a special emphasis on controlling morning blood pressure

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years, insufficiently treated hypertension

Exclusion Criteria:

- Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with essential hypertension
Sampling Method: Non-Probability Sample
Enrollment: 13248 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Changes in morning blood pressure (BP) | Pre-dose, up to 6 months after start of treatment
Changes in metabolic laboratory parameters | Pre-dose, up to 6 months after start of treatment
Changes in morning blood pressure in patients with or without telemonitoring (TM) of BP | Pre-dose, up to 6 months after start of treatment
Investigator assessment of efficacy in reducing morning hypertension on a 5-point rating scale | Up to 6 months after start of treatment
Investigator assessment of effects on metabolism on a 3-point rating scale | Up to 6 months after start of treatment
Investigator assessment of tolerability on a 5-point rating scale | Up to 6 months after start of treatment
Number of patients with adverse events | Up to 6 months
Changes in morning heart rate | Pre-dose, up to 6 months after start of treatment